CLINICAL TRIAL: NCT02374593
Title: Targeted Levothyroxine Dosing in Infants With Congenital Hypothyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erica Eugster (Other)
Responsible Party: Sponsor-Investigator, Erica Eugster, Pediatric Endocrinologist, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1401199401
Record Dates: First submitted 2015-02-18; First posted 2015-03-02 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Congenital Hypothyroidism
MeSH Terms: conditions — Congenital Hypothyroidism | interventions — Thyroxine; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Targeted dosing (Experimental): Patients in this arm will receive targeted levothyroxine dosing based on thyroid anatomy on ultrasound as follows: 10 mcg/kg for normal gland, 12 mcg/kg for ectopic gland, 15 mcg/kg for athyreosis.
  Interventions: Drug: Levothyroxine; Device: Ultrasound

INTERVENTIONS:
Drug: Levothyroxine — Levothyroxine dose will be adjusted at the first clinic visit based on thyroid anatomy on ultrasound.
Device: Ultrasound

SUMMARY:
This is a clinical study comparing targeted levothyroxine dosing based on thyroid anatomy as visualized on ultrasound (normal vs. ectopic/sublingual vs. athyreosis) to empiric levothyroxine dosing in infants with congenital hypothyroidism. Patients enrolled in the study for targeted dosing will be compared to controls obtained by retrospective chart review. The main outcome is to determine if there is a difference in the frequency of over-treatment and under-treatment during the first 6 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Newborns diagnosed with congenital hypothyroidism (CH).
* Newborns with CH who are treated by a pediatric endocrinologist at Riley Hospital for Children or satellite location.
* Newborns with CH who have thyroid imaging performed (thyroid ultrasound or technetium scan) at diagnosis.

Exclusion Criteria:

* Newborns who do not have CH.
* Newborns with CH who have not had thyroid imaging performed at diagnosis.

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Eugster, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Historical Control: Patients in this arm were treated with levothyroxine empirically with an initial dose between 10-15 mcg/kg/day.
Period: Overall Study
Arm/Group | Targeted Dosing | Historical Control
Started | 24 | 44
Completed | 22 | 44
Not Completed | 2 | 0
Not completed — non-compliant | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Targeted Dosing | Historical Control | Total
Number analyzed (Participants) | 22 | 44 | 66
Age, Continuous [Mean (Full Range); unit: weeks] | 1 [0 to 2] | 1 [0 to 2] | 1 [0 to 2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 28 | 42
  Male | 8 | 16 | 24
Region of Enrollment [Number; unit: participants]
  United States | 22 | 44 | 66

OUTCOME MEASURES:

1. Primary Outcome: Dose Adjustments
Description: Thyroid labs (TSH and fT4/T4) will be monitored per standard care: 2 weeks after initiation of levothyroxine and once monthly during the first 6 months of treatment. The number of dose adjustments required per participant during the first 6 months of treatment were recorded.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Number of dose adjustments
Arm/Group | Targeted Dosing | Historical Control
Number analyzed (Participants) | 22 | 44
Number of dose adjustments | 2.5 (0.334) | 2.4 (0.211)

2. Secondary Outcome: Number of Adjustments Due to Overtreatment in Subjects With Athyreosis, Ectopic and Eutopic Thyroid Glands Compared With Controls
Description: Whether the dose adjustment was made for overtreatment was noted as based on TSH and fT4/T4 results
Time Frame: 6 months
Measure: Mean (Standard Error); unit: dose adjustments
Groups:
- Patients With Athyreosis: Patients in this arm will receive targeted levothyroxine dosing based on thyroid anatomy at 15 mcg/kg for athyreosis.
  Levothyroxine: Levothyroxine dose will be adjusted at the first clinic visit based on thyroid anatomy on ultrasound.
  Ultrasound
- Patients With Dysgenetic Thyroids: patients with dysgenetic thyroids
- Patients With Eutopic Thyroids: patients with eutopic thyroids
- Historical Controls: see title
Arm/Group | Patients With Athyreosis | Patients With Dysgenetic Thyroids | Patients With Eutopic Thyroids | Historical Controls
Number analyzed (Participants) | 10 | 4 | 8 | 44
dose adjustments | 2.7 (0.275) | 2 (0.275) | 1 (0.275) | 2 (0.275)

ADVERSE EVENTS:
Description: Adverse events were not monitored as all subjects were treated according to existing clinical standards of care
Arm/Group | Targeted Dosing | Historical Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes